CLINICAL TRIAL: NCT03233282
Title: Electrophysiological and Bioenergetic Study of Variations in Cognitive and Physical Performance in Healthy Humans: EEG Monitoring for PERFormance Anticipation
Brief Title: EEG Monitoring for PERFormance Anticipation
Acronym: MEEGAPERF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL16_0661
Record Dates: First submitted 2017-04-25; First posted 2017-07-28 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Healthy
MeSH Terms: interventions — Magnetoencephalography; Oxygen Consumption

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cognitive Fatigability (Other)
  Interventions: Other: Electroencephalography (EEG) multi-sensor; Other: Magnetoencephalography (MEG); Other: Behavioral Measures; Other: Reaction time measurement; Other: Assessment of physical performance; Other: Electrooculogram (EOG); Other: Electromyogram (EMG); Other: Electrocardiogram with 3 leads
- Physical Fatigability (Other)
  Interventions: Other: Electroencephalography (EEG) multi-sensor; Other: Magnetoencephalography (MEG); Other: Behavioral Measures; Other: Reaction time measurement; Other: Assessment of physical performance; Other: Electrooculogram (EOG); Other: Electromyogram (EMG); Other: Electrocardiogram with 3 leads; Other: Electrodermogram (EDG); Other: Consumption of O2 (VO2); Other: Production of CO2 (VCO2)

INTERVENTIONS:
Other: Electroencephalography (EEG) multi-sensor — Electrophysiological measurements of cerebral activity will be performed by multi-sensor electroencephalography (EEG), which is a non-invasive method.
Other: Magnetoencephalography (MEG) — Electrophysiological measurements of brain activity will be performed by magnetoencephalography (MEG) which is a non-invasive method.
Other: Behavioral Measures — The evaluation of cognitive performance will be carried out by means of behavioral measures, push-button type, handling of a mouse or a joystick.
Other: Reaction time measurement — The assessment of cognitive performance will be carried out using standard behavioral measures, such as reaction time measurement.
Other: Assessment of physical performance — The assessment of physical performance will be based both on bioenergetic measurements and on quantitative data collected in continuous and relative to the effort (eg instantaneous pedaling speed).
Other: Electrooculogram (EOG) — In order to extract artifacts and verify the physical performances of the subjects, under the conditions of physical fatigability, peripheral electrophysiological recordings will be necessary and complementary to meet the objectives set in this study.
Other: Electromyogram (EMG) — In order to extract artifacts and verify the physical performances of the subjects, under the conditions of physical fatigability, peripheral electrophysiological recordings will be necessary and complementary to meet the objectives set in this study.
Other: Electrocardiogram with 3 leads — In order to extract artifacts and verify the physical performances of the subjects, under the conditions of physical fatigability, peripheral electrophysiological recordings will be necessary and complementary to meet the objectives set in this study.
Other: Electrodermogram (EDG) — In order to extract artifacts and verify the physical performances of the subjects, under the conditions of physical fatigability, peripheral electrophysiological recordings will be necessary and complementary to meet the objectives set in this study.
  Arms: Physical Fatigability
Other: Consumption of O2 (VO2) — In order to extract artifacts and verify the physical performances of the subjects, under the conditions of physical fatigability, peripheral electrophysiological recordings will be necessary and complementary to meet the objectives set in this study.
  Arms: Physical Fatigability
Other: Production of CO2 (VCO2) — In order to extract artifacts and verify the physical performances of the subjects, under the conditions of physical fatigability, peripheral electrophysiological recordings will be necessary and complementary to meet the objectives set in this study.
  Arms: Physical Fatigability

SUMMARY:
Identify, characterize and then validate electrophysiological markers linking electrophysiological cerebral activity and performance in cognitive and physical fatigability in humans. To do this, noninvasive explorations of electroencephalography (EEG) and magnetoencephalography (MEG) will be carried out under two conditions of different experiments, the first one that induces a cognitive fatigability and the second one that induces physical fatigability.

ELIGIBILITY:
Inclusion Criteria MGPFco group:

* Adult subjects, male or female, right-handed or left-handed, from 18 years up to 70 years;
* Having duly completed the entire confidential medical questionnaire;
* Written consent of free, informed and express participation;
* No hearing problems;
* Having normal or corrected vision;
* Affiliation to a Social Security scheme.

Inclusion Criteria MGPFph group:

* Adult subjects, male or female, right-handed or left-handed, from 18 years up to 35 years;
* Practicing at least five hours of sports per week;
* Presenting a certificate of no contraindication to an exercise test, intense sports practice or an energy sport in competition of the current year;
* Having duly completed the entire confidential medical questionnaire;
* Without cardiovascular or motor disability;
* Without tumoral, inflammatory, cardiac, pulmonary, renal, digestive (malabsorption syndrome) or liver disease;
* Written consent of free, informed and express participation;
* Affiliation to a Social Security scheme.

Exclusion Criteria:

* Pregnant women, nursing mothers or those of childbearing age without contraception
* Persons under guardianship, curatorship or any other administrative or judicial measure of deprivation of liberty or of liberty
* Persons protected by the law
* Persons who have performed a maximum stress test within 15 days of the date of inclusion,
* In the course of drug treatments against indicated for the protocol (treatment for neurological diseases, psychiatric ...).
* Metal implants incompatible with MRI (for the subjects concerned, see appendices)
* Metallic implants incompatible with the MEG (for the subjects concerned, see appendices)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2013-05-30 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Identify electrophysiological markers in humans depending on whether the experimental conditions induce cognitive fatigability. | 7 hours
  The evaluation of cognitive performance will be carried out by means of conventional behavioral measures, of the press-button type, handling of a mouse or of a joystick and measurement of reaction time.
Identify electrophysiological markers in humans depending on whether the experimental conditions induce physical fatigability with EEG. | 7 hours
  Electrophysiological measurements of cerebral activity will be performed by multi-sensor electroencephalography (EEG).
Identify electrophysiological markers in humans depending on whether the experimental conditions induce physical fatigability with MEG. | 7 hours
  Electrophysiological measurements of cerebral activity will be carried out by magnetoencephalography (MEG)

SECONDARY OUTCOMES:
Refine (locate at the level of the cortex), the origin of these physiological markers | 7 hours
  Several types of recordings, passive and non-invasive, will be realized:
  * Electrooculogram (EOG);
  * electromyography (EMG);
  * electrocardiogram (ECG); Systematically in "physical" experiments and for some "cognitive" experiments.
Distinguish between different time scales of performance | 7 hours
  Several types of recordings, passive and non-invasive, will be realized:
  * electrodermogram (EDG);
  * the consumption of O2 (VO2);
  * production of CO2 (VCO2). Only and systematically, in "physical" experiments.

CONTACTS AND LOCATIONS:
Overall Officials: Julien JUNG, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, HFME, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poinsard L, Berthomier C, Clemencon M, Brandewinder M, Essid S, Damon C, Rigaud F, Benichoux A, Maby E, Fornoni L, Bouchet P, Beers PV, Massot B, Revol P, Creveaux T, Collet C, Mattout J, Pialoux V, Billat V. EEG-Metabolic Coupling and Time Limit at V O2max During Constant-Load Exercise. J Funct Morphol Kinesiol. 2025 Sep 26;10(4):369. doi: 10.3390/jfmk10040369. PMID 41133559
- [Background] Véronique Billat, Christian Berthomier, Michel Clémençon, Marie Brandewinder, Slim Essid, Cécilia Damon, François Rigaud, Alexis Bénichoux, Emmanuel Maby, Lesly Fornoni, Patrick Bouchet , Pascal Van Beers, Bertrand Massot, Patrice Revol, Luc Poinsard, Thomas Creveaux, Christian Collet, Jérémie Mattout and Vincent Pialoux. Electroencephalography Response during an Incremental Test According to the VO2max Plateau Incidence. Applied Sciences. 2024, 14, 5411.
- [Derived] Seguin P, Maby E, Fouillen M, Otman A, Luaute J, Giraux P, Morlet D, Mattout J. The challenge of controlling an auditory BCI in the case of severe motor disability. J Neuroeng Rehabil. 2024 Jan 18;21(1):9. doi: 10.1186/s12984-023-01289-3. PMID 38238759